CLINICAL TRIAL: NCT04748653
Title: Comprehensive Reintegration Assistance for Women With Obstetric Fistula
Brief Title: Fistula Reintegration Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Makerere University (Other); Mama, LLC (Unknown); Mulago Hospital, Uganda (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P0527552; R00HD086232 (NIH)
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Female Genital Fistula; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: The intervention incorporates 15 health education sessions, 6 psychosocial counseling sessions, 15 physiotherapy sessions, and an economic investment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-component reintegration intervention (Experimental): There is one arm for the feasibility and acceptability study - all intervention participants will receive the intervention: health education, psychosocial counseling, physiotherapy, and economic investment.
  Interventions: Behavioral: Multi-component reintegration intervention

INTERVENTIONS:
Behavioral: Multi-component reintegration intervention — The intervention incorporates health education, psychosocial counseling, physiotherapy and economic investment.

SUMMARY:
This is a pilot study to test the feasibility and acceptability of a multi-component facility-based intervention designed to be provided adjunct to genital fistula surgery incorporating: health education, psychosocial counseling, physiotherapy, and economic investment. We will include a total of 30 women in the study, and follow them for 6-months using a mixed-methods strategy for feasibility and acceptability assessment.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery for female genital fistula
* Age 18 or above, or emancipated minor per Ugandan law

Exclusion Criteria:

* No further criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison El Ayadi, ScD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Mulago Specialized Women's and Children's Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multi-component Reintegration Intervention
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Multi-component Reintegration Intervention
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.5 [24.5 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Planned Intervention Sessions That Were Delivered
Description: Number of planned intervention session over the total number of planned interention sessions
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of planned sessions
Arm/Group | Multi-component Reintegration Intervention
Number analyzed (Participants) | 12
percentage of planned sessions | 96.2 [95 to 97.5]

2. Primary Outcome: Number of Participants Reporting to be "Satisfied" or "Very Satisfied" About Their Overall Experience With the Intervention on a Five-point Likert Scale at Six Weeks Over the Total Number of Intervention Participants.
Description: Number of participants reporting to be "satisfied" or "very satisfied" about their overall experience participating in the intervention on a five-point Likert scale at six weeks over the total number of participants.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-component Reintegration Intervention
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Change in Reintegration Score
Description: Mean change in reintegration score from pre-intervention (baseline) to post (6 months) on the post-fistula repair reintegration instrument (range 0-100, higher indicating better)
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Multi-component Reintegration Intervention
Number analyzed (Participants) | 12
scores on a scale | 30.5 [23.5 to 39.5]

4. Secondary Outcome: Number of Participants Reporting to be "Satisfied" or "Very Satisfied" About Their Experience With the Health Education Component of the Intervention on a Five-point Likert Scale at Six Weeks Over the Total Number of Intervention Participants
Description: Number of participants reporting to be "satisfied" or "very satisfied" about their experience participating in the health education component of the intervention on a five-point Likert scale at six weeks over the total number of participants.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-component Reintegration Intervention
Number analyzed (Participants) | 12
Participants | 12

5. Secondary Outcome: Number of Participants Reporting to be "Satisfied" or "Very Satisfied" About Their Experience Participating in the Psychosocial Counseling Component of the Intervention on a Five-point Likert Scale at Six Weeks Over the Total Number of Participants.
Description: Number of participants reporting to be "satisfied" or "very satisfied" about their experience participating in the psychosocial counseling component of the intervention on a five-point Likert scale at six weeks over the total number of participants.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-component Reintegration Intervention
Number analyzed (Participants) | 12
Participants | 12

6. Secondary Outcome: Number of Participants Reporting to be "Satisfied" or "Very Satisfied" About Their Experience With the Physiotherapy Component of the Intervention on a Five-point Likert Scale at Six Weeks Over the Total Number of Intervention Participants.
Description: Number of participants reporting to be "satisfied" or "very satisfied" about their experience with the physiotherapy component of the intervention on a five-point Likert scale at six weeks over the total number of intervention participants.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-component Reintegration Intervention
Number analyzed (Participants) | 12
Participants | 12

7. Secondary Outcome: Number of Participants Reporting to be "Satisfied" or "Very Satisfied" About Their Experience With the Economic Empowerment Component of the Intervention on a Five-point Likert Scale at Six Weeks Over the Total Number of Intervention Participants
Description: Number of Participants Reporting to be "Satisfied" or "Very Satisfied" About Their Experience With the Economic Empowerment Component of the Intervention on a Five-point Likert Scale at Six Weeks Over the Total Number of Intervention Participants
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-component Reintegration Intervention
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Multi-component Reintegration Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT04748653/Prot_SAP_ICF_000.pdf